CLINICAL TRIAL: NCT03329651
Title: The Interaction Between Metformin and Acute Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kristian Karstoft (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Kristian Karstoft, Principal Investigator, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: H-17012307-1
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Impaired Glucose Tolerance; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin treatment (Experimental)
  Interventions: Drug: Metformin treatment
- Placebo treatment (Placebo Comparator)
  Interventions: Drug: Placebo treatment

INTERVENTIONS:
Drug: Metformin treatment — Daily treatment with metformin tablets for 24 days according to the following scheme:
  Day 1-4: Metformin tablet 500 mg x 2 Day 5-8: Metformin tablet 1000 + 500 mg Day 9-24: Metformin tablet 1000 mg x 2
  Arms: Metformin treatment
Drug: Placebo treatment — Daily treatment with placebo tablets for 24 days according to the following scheme:
  Day 1-4: Placebo tablet 500 mg x 2 Day 5-8: Placebo tablet 1000 + 500 mg Day 9-24: Placebo tablet 1000 mg x 2
  Arms: Placebo treatment

SUMMARY:
Physical activity is a first line treatment for patients with type 2 diabetes (T2D), however, the vast majority of patients with T2D do not achieve satisfying glycemic control with physical activity alone, which is why pharmacological treatment with metformin is most often initiated.

It is known that metformin and exercise both activates 5' adenosine monophosphate-activated protein kinase (AMPK) in skeletal muscle and liver, and the activation of AMPK results in many different metabolic effects, including improvements in glycemic control. Because of this similarity in mechanism of action, an interaction between metformin and exercise is plausible, but knowledge in the area is sparse. Thus, the aim of this study is to assess the effects of acute physical activity with and without concomitant metformin treatment, in order to investigate whether an interaction between the two occur.

Subjects with impaired glucose tolerance will be randomized (1:1) to metformin/placebo treatment in a double-blinded way. Following a treatment run-in period of 17 days, two experimental days (one with acute exercise and one without acute exercise), separated by one week, will be performed in each subject.

This registration concerns a sub-study of another study which has previously been registrered at ClinicalTrials.gov (Unique Protocol ID: H-17012307). The specific outcomes in this registration have not previously been registered.

ELIGIBILITY:
Inclusion Criteria:

* Glucose-lowering-medication naïve T2D and/or subjects with impaired glucose tolerance defined as: 2-h plasma glucose (PG) in the 75-g OGTT (7.8-11.0 mmol/L) and/or HbA1c (39-47 mmol/mol)
* Caucasian
* BMI > 25 but < 40 kg/m2
* Low to moderate physically active (≤90 min of structured physical activity/week)

Exclusion Criteria:

* Pregnancy
* Smoking
* Glucose-lowering treatment
* Treatment with steroids and other immunomodulating drugs
* Contraindication to increased levels of physical activity
* Liver disease (ALAT elevated more than 3 times above upper normal limit, or reduced levels of the liver function markers albumin and KF II+VII+X)
* Renal insufficiency (eGFR<60 ml/min)
* Prior history of lactic acidosis
* HbA1c >55 mmol/mol and/or 2-hPG in the 75-g OGTT > 15 mmol/L

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Difference in postprandial glycemic control as assessed by mean blood glucose concentration during a 4 hour mixed-meal tolerance test | Day 17 (no acute exercise [control day]) and 24 (following an acute exercise bout)

SECONDARY OUTCOMES:
Difference in endogenous glucose production as assessed by rate of infused glucose tracer appearance in blood | Day 17 (no acute exercise [control day]) and 24 (following an acute exercise bout)
Difference in exogenous glucose uptake as assessed by rate of ingested glucose tracer appearance in blood | Day 17 (no acute exercise [control day]) and 24 (following an acute exercise bout)
Difference in peripheral glucose uptake as assessed by rate of glucose disappearance from blood | Day 17 (no acute exercise [control day]) and 24 (following an acute exercise bout)

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Karstoft, MD, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Center for aktiv sundhed, Copenhagen, Copenhagen N, Denmark

IPD SHARING:
Plan to Share IPD: Undecided